CLINICAL TRIAL: NCT00993616
Title: A Phase II Evaluation of Belinostat (NSC #726630) and Carboplatin (NSC #241240) in the Treatment of Recurrent or Persistent Platinum-Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Belinostat and Carboplatin in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer That Did Not Respond to Carboplatin or Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-01663; NCI-2010-01663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000656707; GOG-0126T (Other: Gynecologic Oncology Group); GOG-0126T (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2014-01-21 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Brenner Tumor; Fallopian Tube Cancer; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mixed Epithelial Carcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Adenocarcinoma; Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — belinostat; Carboplatin

ARMS (1):
- Treatment (Experimental): Patients receive belinostat IV over 30 minutes on days 1-5 and carboplatin IV over 30-60 minutes on day 3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who are clinically responding or who, in the opinion of their physician, would continue to benefit from treatment may continue treatment beyond 6 courses.
  Interventions: Drug: belinostat; Drug: carboplatin

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin

SUMMARY:
This phase II trial is studying how well giving belinostat together with carboplatin works in treating patients with recurrent or persistent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer that did not respond to carboplatin or cisplatin. Belinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving belinostat together with carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the antitumor activity of belinostat and carboplatin in patients with persistent or recurrent platinum-resistant ovarian, fallopian tube, or primary peritoneal cancer, measured by objective response rate and the frequency of progression- free survival at 6 months.

II. To determine the nature and degree of toxicity of belinostat in combination with carboplatin in this cohort of patients.

OUTLINE: This is a multicenter study.

Patients receive belinostat IV over 30 minutes on days 1-5 and carboplatin IV over 30-60 minutes on day 3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who are clinically responding or who, in the opinion of their physician, would continue to benefit from treatment may continue treatment beyond 6 courses.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* Patients with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.)
* All patients must have measurable disease as defined by RECIST 1.1; measureable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority GOG protocol, if one exists; in general, this would refer to any active GOG Phase III or Rare Tumor protocol for the same patient population
* Patients must have a GOG Performance Status of 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated UTI)
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included non-cytotoxic therapy, intraperitoneal therapy, high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
* Patients must be considered platinum resistant or refractory according to the following criteria:

  * Patients must have had progression of disease on or within 6 months of their last platinum dose
  * Progression of disease is defined according to RECIST 1.1
  * The development of CA125 elevation on or within 6 months of last platinum treatment, in the absence of radiographic progression according to RECIST 1.1, is not considered platinum resistance for the purposes of this study
* Patients who have NOT received prior therapy with taxane-based chemotherapy MUST receive a second regimen that includes paclitaxel or docetaxel
* Patients must be considered paclitaxel-resistant, i.e., have had a treatment-free interval following paclitaxel of less than six months, or have progressed during paclitaxel-based therapy
* Patients must have NOT received any additional cytotoxic chemotherapy for management of recurrent or persistent disease, including retreatment with initial chemotherapy regimens except as noted above; (note: Optimal evaluation of the safety and efficacy of new chemotherapy regimens is best performed in patients with minimal prior therapy; non-investigational therapy, such as retreatment with platinum and/or paclitaxel, is non-curative in the setting of recurrent disease, and can generally be safely administered to patients following participation in a phase II trial)
* Patients are allowed to receive, but are not required to receive, one additional non-cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Non-cytotoxic (biologic or cytostatic) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to the NCI Common Terminology Criteria (CTCAE v3.0) grade 1
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), per CTCAE v.3.0 grade 1
* Bilirubin less than or equal to 1.5 x ULN (CTCAE v.3.0 grade 1)
* SGOT (AST) less than or equal to 3 x ULN (per the CTCAE v.3.0 grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v.3.0 grade 1)
* Neuropathy (sensory and motor) less than or equal to the CTCAE v3.0 grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had prior therapy with Belinostat (PXD101) or other HDAC inhibitors
* Patients who have received radiation to more than 25% of marrow-bearing areas
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, and other specific malignancies as noted below, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian cancer are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian cancer are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients must not use concomitant medications on PXD infusion days that may cause Torsade de Pointes; medications associated with this risk include:

  * Amiodarone, Arsenic trioxide, Bepridil, Cisapride, Disopyramide, Dofetilide, Droperidol, Erythromycin, Felbamate, Flecainide, Fluoxetine, Halofantrine, Haloperidol, Ibutilide, Levofloxacin, Mesoridazine, Pentamidine, Procainamide, Quinidine, Sotalol, Sparfloxacin, or Thioridazine
* Patients with significant cardiovascular disease defined as:

  * Unstable angina pectoris, uncontrolled hypertension (blood pressure > 150/90 despite maximal medical therapy), congestive heart failure related to primary cardiac disease, any condition requiring anti-arrhythmic therapy, ischemic or severe valvular heart disease, or history of myocardial infarction within 6 months of trial entry
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Dizon, Principal Investigator — Gynecologic Oncology Group
Locations (81):
- United States (81):
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 29
Completed | 27 (Number of eligible and evaluable participants)
Not Completed | 2
Not completed — No tumor at entry | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Number of eligible and evaluable participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (6.8)
Age, Customized [Number; unit: participants]
  40-49 years | 2
  50-59 years | 8
  60-69 years | 15
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 1
  Clear Cell Carcinoma | 2
  Mixed Epithelial Carcinoma | 1
  Serous Adenocarcinoma | 23

OUTCOME MEASURES:

1. Primary Outcome: Objective Response by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (Version 1.1)
Description: Per Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (version 1.1): Complete Response (CR) is disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Increasing Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions); Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest
Time Frame: From study entry, up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
participants
  Complete Response | 1
  Increase Disease | 8
  Partial Response | 1
  Stable Disease | 12
  Indeterminate | 5

2. Primary Outcome: Frequency and Severity of Observed Adverse Effects Graded According to NCI CTCAE Version 3.0
Time Frame: Every cycle during treatment and 30 days after the end of treatment
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1: Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2: Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3: Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4: Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5: Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Participants
  Leukopenia | 12 | 5 | 9 | 1 | 0 | 0
  Thrombocytopenia | 14 | 5 | 4 | 2 | 2 | 0
  Neutropenia | 13 | 2 | 6 | 4 | 2 | 0
  Anemia | 6 | 10 | 9 | 2 | 0 | 0
  Other hematologic | 26 | 1 | 0 | 0 | 0 | 0
  Allergy/immunology | 23 | 0 | 2 | 1 | 1 | 0
  Auditory/ear | 26 | 0 | 1 | 0 | 0 | 0
  Cardiac | 26 | 1 | 0 | 0 | 0 | 0
  Coagulation | 25 | 1 | 1 | 0 | 0 | 0
  Constitutional | 10 | 10 | 6 | 1 | 0 | 0
  Dermatologic | 22 | 3 | 2 | 0 | 0 | 0
  Endocrine | 26 | 1 | 0 | 0 | 0 | 0
  Nausea | 6 | 14 | 5 | 2 | 0 | 0
  Vomiting | 14 | 9 | 1 | 3 | 0 | 0
  Gastrointestinal | 10 | 8 | 7 | 2 | 0 | 0
  Genitourinary/renal | 26 | 1 | 0 | 0 | 0 | 0
  Hemorrhage | 25 | 1 | 0 | 0 | 0 | 1
  Lymphatics | 26 | 1 | 0 | 0 | 0 | 0
  Metabolic | 17 | 7 | 1 | 2 | 0 | 0
  Musculoskeletal | 25 | 2 | 0 | 0 | 0 | 0
  Neurosensory | 21 | 5 | 1 | 0 | 0 | 0
  Other neurological | 22 | 3 | 2 | 0 | 0 | 0
  Ocular/visual | 26 | 1 | 0 | 0 | 0 | 0
  Pain | 15 | 8 | 4 | 0 | 0 | 0
  Pulmonary | 21 | 6 | 0 | 0 | 0 | 0
  Vascular | 25 | 0 | 2 | 0 | 0 | 0

3. Primary Outcome: Progression Free Survival at 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: Every other cycle for 6 months
Population: Eligible and treated patients
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
percentage of participants | 29.6

4. Other Pre Specified Outcome: Duration of Progression-free Interval for All Patients
Time Frame: up to 5 years
Population: Please note: this outcome measure is not an endpoint as per the protocol document. Data will not be reported.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From study entry up to 5 years
Description: From the period of protocol activation through September 30, 2011, Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (CTCAE v3.0) are utilized. (9/26/11) Beginning October 1, 2011, the NCI Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 will be utilized.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 9/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=27)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Obstruction, Gastrointestinal - Small Bowel Not otherwise specified (Gastrointestinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 1
Hemorrhage, Gastrointestinal - Upper Gastrointestinal Not Otherwise Specified (Vascular disorders) | 1
Infection with normal or Grade 1 Or 2 Absolute neutrophil count: Blood (Infections and infestations) | 1
Somnolence (Nervous system disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=27)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 3
Neutrophils (Blood and lymphatic system disorders) | 15
Platelets (Blood and lymphatic system disorders) | 12
Leukocytes (Blood and lymphatic system disorders) | 15
Hemoglobin (Blood and lymphatic system disorders) | 21
Palpitations (Cardiac disorders) | 2
Partial thromboplastin time (Vascular disorders) | 2
Weight Gain (General disorders) | 2
Fatigue (General disorders) | 18
Insomnia (General disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 4
Hot Flashes (Endocrine disorders) | 4
Distention (Gastrointestinal disorders) | 2
Mucositis (Functional/Symptomatic) - Oral Cavity (Gastrointestinal disorders) | 2
Obstruction, Gastrointestinal - Small Bowel Not otherwise specified (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 6
Creatinine (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 4
Neuropathy-Sensory (Nervous system disorders) | 11
Blurred Vision (Eye disorders) | 2
Pain: Head/Headache (General disorders) | 6
Pain: Abdominal Pain Not otherwise specified (General disorders) | 7
Pain: Muscle (General disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less